CLINICAL TRIAL: NCT02041156
Title: Long-term Effects of Basic Aerobic Training Combined With Either Resistance - or Balance Training in CKD Patients - a Comparative Study
Brief Title: Effects of Different Exercise Training Programs in CKD 4-5
Acronym: RENEXC
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Region Skane (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2011:369
Record Dates: First submitted 2014-01-07; First posted 2014-01-20 (Estimated); Last update posted 2016-09-23 (Estimated); Status verified 2016-09

CONDITIONS: Chronic Kidney Disease
MeSH Terms: conditions — Renal Insufficiency, Chronic | interventions — Resistance Training

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- aerobic with resistance training (Experimental): Regular aerobic activity combined with 3 sessions/week of resistance training totalling 150 minutes per week of physical activity
  Interventions: Other: aerobic and resistance training
- aerobic with balance training (Active Comparator): Regular aerobic activity combined with 3 sessions/week of balance training totalling 150 minutes per week of physical activity
  Interventions: Other: aerobic combined with balance training

INTERVENTIONS:
Other: aerobic and resistance training
  Arms: aerobic with resistance training
Other: aerobic combined with balance training
  Arms: aerobic with balance training

SUMMARY:
The investigators' purpose is to study which exercise training modality: aerobic physical activity in conjunction with either resistance training or balance training, is most beneficial in patients with chronic kidney disease (CKD 4-5: GFR < 30 ml/min/1.73mUP[2]). Furthermore, our purpose is to evaluate the long-term effects of exercise training on functional status, cardiovascular morbidity, blood pressure control, heart rate variability, cardiac function, inflammation, body composition, nutritional status, progression of uraemia and health related quality of life. This interventional study is prospective, randomized and controlled comprising 150 prevalent and incident patients from our outpatient clinic. Patients are invited to participate in the study consecutively, irrespective of basic functional status. At start patients are randomised either to resistance or balance training and the programme is adapted and individualised to each patient's actual physical status and ability. The exercise prescription is to exercise for 30 minutes/day, 5 days/week, keeping the intensity constant at a level of "somewhat strenuous" to "strenuous" on the Borg scale rate of perceived exertion. The total observation period is 12 months with checks every four months. Although exercise training is a recommended therapy in CKD, there is a lack of medical and scientific evidence on optimal prescription. We hope that this study will provide evidence-based knowledge on exercise prescription and its effects on various risk factors in CKD patients. Finally, if patients achieve a higher degree of physical functional capacity they should be able to maintain an autonomous lifestyle, resulting in considerable reductions in societal costs for care and transportation.

ELIGIBILITY:
Inclusion Criteria:

* CKD 4 and 5
* over 18 years of age
* no neurological or orthopedic impairments
* stable cardiac status

Exclusion Criteria:

* not on renal replacement therapy
* no severe electrolyte disturbances

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2011-10; Primary Completion 2017-02 (Estimated); Study Completion 2017-02 (Estimated)

PRIMARY OUTCOMES:
Physical function | 4, 8 and 12 months
  6 minutes walking test, 30 seconds sit to stand, stair climbing, handgrip strength, Isometric quadriceps strength, functional reach, standing heel rise, toes lift, picking-up test, Berg balance scale

SECONDARY OUTCOMES:
Cardiovascular morbidity | after 12 months
Body composition | after 12 months
Quality of Life | 4,8 and 12 months
Inflammatory activity | 4, 8 and 12 months
Bone density | 12 months

OTHER OUTCOMES:
Compliance to exercise training protocol | 4, 8 and 12 month

CONTACTS AND LOCATIONS:
Overall Officials: Naomi Clyne, MD, PhD, Study Director — Lund University; Matthias Hellberg, MD, Principal Investigator — Lund University
Locations (1):
- Skåne University Hospital, Lund, Sweden

REFERENCES:
- [Derived] Petrauskiene V, Hellberg M, Svensson P, Clyne N. Markers of bone turnover after 12 months of exercise in patients with chronic kidney disease 3-5: a post-hoc analysis of RENEXC - a randomized controlled trial. BMC Nephrol. 2025 Oct 13;26(1):561. doi: 10.1186/s12882-025-04501-9. PMID 41083942
- [Derived] Denguir S, Hellberg M, Almquist M, Clyne N. Survival in patients with CKD 3-5 after 12 months of exercise training - a post-hoc analysis of the RENEXC trial. BMC Nephrol. 2025 Jan 23;26(1):36. doi: 10.1186/s12882-024-03915-1. PMID 39849350
- [Derived] Zhou Y, Hellberg M, Hellmark T, Hoglund P, Clyne N. Twelve months of exercise training did not halt abdominal aortic calcification in patients with CKD - a sub-study of RENEXC-a randomized controlled trial. BMC Nephrol. 2020 Jun 22;21(1):233. doi: 10.1186/s12882-020-01881-y. PMID 32571327
- [Derived] Zhou Y, Hellberg M, Hellmark T, Hoglund P, Clyne N. Muscle mass and plasma myostatin after exercise training: a substudy of Renal Exercise (RENEXC)-a randomized controlled trial. Nephrol Dial Transplant. 2021 Jan 1;36(1):95-103. doi: 10.1093/ndt/gfz210. PMID 31848626